CLINICAL TRIAL: NCT05960708
Title: A Randomized, Double-Blind, Placebo/Active Controlled, Single Dose, Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Following Subcutaneous Injections of YH35324 in Patients with Various Allergic Diseases
Brief Title: A Single Dose, Phase 1 Study of YH35324 in Patients with Various Allergic Diseases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YH35324-103
Record Dates: First submitted 2023-07-13; First posted 2023-07-27 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Allergic Disease; Chronic Spontaneous Urticaria; Chronic Inducible Urticaria; Cold Urticaria
Keywords: GI-301; YH35324; Allergic disease; CSU; CINDU; Cold urticaria
MeSH Terms: conditions — Chronic Urticaria; Chronic Inducible Urticaria; Cold Urticaria | interventions — Omalizumab; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each IP will be labeled with a unique IP number, and the number will be associated with the randomized treatment group. Interactive Web Response System (IWRS) will be used to assign a randomization number and IP number.
  As YH35324, placebo, and omalizumab differ in appearance, the assigned treatment group of subjects should be disclosed to study pharmacists and unblinded staff who prepare (taking an appropriate and correct amount (mL) of the IP based on the subject's body weight into a syringe), dispense, and administer the IPs, in order to maintain the blind. Therefore, the treatment group information of subjects will be checked through IWRS with limited access before administration of the IP, and only study pharmacists and unblinded staff are allowed to access the system.
  The study pharmacists and unblinded staff should not disclose the assigned treatment group of enrolled subjects to the principal investigator or study staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- YH35324 (Experimental): [Part 1] A total of 18 subjects will be randomized in a 1:1:1 ratio to the YH35324 A mg/kg, YH35324 B mg/kg, or omalizumab group.
  [Part 2] A total of 9 subjects will be randomized in a 2:1 ratio to the YH35324 B mg/kg or placebo group.
  [Part 3] A total of 9 subjects will be randomized in a 2:1 ratio to the YH35324 B mg/kg or placebo group.
  Interventions: Drug: YH35324
- Omalizumab (Active Comparator): [Part 1] A total of 18 subjects will be randomized in a 1:1:1 ratio to the YH35324 A mg/kg, YH35324 B mg/kg, or omalizumab group.
  Interventions: Drug: Omalizumab
- Placebo (Placebo Comparator): [Part 2] A total of 9 subjects will be randomized in a 2:1 ratio to the YH35324 B mg/kg or placebo group.
  [Part 3] A total of 9 subjects will be randomized in a 2:1 ratio to the YH35324 B mg/kg or placebo group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YH35324 — Subcutaneous injection of YH35324
  Arms: YH35324
Drug: Omalizumab — Subcutaneous injection of Omalizumab
  Other Names: Xolair® prefilled syringe 150 for injection
  Arms: Omalizumab
Drug: Placebo — Subcutaneous injection of None of active ingredient
  Arms: Placebo

SUMMARY:
This study aims to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) following a single subcutaneous injection of YH35324 in subjects with various allergic diseases.

DETAILED DESCRIPTION:
This drug(YH35324) is currently under development as a novel therapeutic agent for various IgE-mediated allergic diseases. Since YH35324 exhibits high binding affinity to human IgE, it prevents serum IgE from binding to receptors on mast cells and basophils, thereby inhibiting histamine release via degranulation following allergen exposures. In addition, YH35324 suppresses autoantibody-dependent effector cell activation by blocking anti-FcεRIα autoantibodies. This study aims to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) following a single subcutaneous injection of YH35324 in subjects with various allergic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged ≥ 19 to ≤ 75 years

[Parts 1 and 2 only]

* Diagnosis of CSU

[Part 2 only]

* Experience of inadequately uncontrolled CSU despite use of omalizumab

[Part 3 only]

* Diagnosis of chronic inducible urticaria (cold urticaria)

Exclusion Criteria:

* History of malignancy within 5 years from screening
* Aspartate transaminase (AST) or alanine transaminase (ALT) level > 2 X the upper limit of normal

[Parts 1 and 2 only]

* Chronic urticaria with clear etiology other than CSU

[Part 3 only]

* Chronic urticaria other than studied chronic inducible urticaria (cold urticaria)

The above information is not intended to contain all considerations relevant to a patient potential participation in a clinical trial.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Occurrence and severity of adverse events (AEs) | Occurrence and severity of adverse events will be observed for 57 days after administration
  To evaluate the safety and tolerability following single administration of YH35324

SECONDARY OUTCOMES:
Change in serum free IgE level | Change in serum free IgE will be observed for 57 days after administration
  To evaluate the PD profile on serum IgE following single administration of YH35324

OTHER OUTCOMES:
Maximum Serum Concentration(Cmax) | Serum concentrations of YH35324 will be observed for 57 days after administration
  To evaluate the PK profile following single administration of YH35324
Area Under the Serum Concentration-Time Curve from Zero to the Time of the Last Quantitative Concentration (AUClast) | Serum concentrations of YH35324 will be observed for 57 days after administration
  To evaluate the PK profile following single administration of YH35324
Area Under the Serum Concentration-Time Curve from Zero to Infinity (AUCinf) | Serum concentrations of YH35324 will be observed for 57 days after administration
  To evaluate the PK profile following single administration of YH35324
Time to Maximum Serum Concentration (Tmax) | Serum concentrations of YH35324 will be observed for 57 days after administration
  To evaluate the PK profile following single administration of YH35324
Terminal Elimination Rate Constant, Apparent Terminal Elimination Half-life (t1/2) | Serum concentrations of YH35324 will be observed for 57 days after administration
  To evaluate the PK profile following single administration of YH35324
Apparent Serum Clearance (CL/F) | Serum concentrations of YH35324 will be observed for 57 days after administration
  To evaluate the PK profile following single administration of YH35324
Apparent Volume of Distribution (Vz/F) | Serum concentrations of YH35324 will be observed for 57 days after administration
  To evaluate the PK profile following single administration of YH35324
Change in serum total IgE level | Change in serum total IgE will be observed for 57 days after administration
  To evaluate the exploratory PD profile following single administration of YH35324
Change in FcƐRI expression on basophil surface | Change in FcƐRI expression on basophil surface will be observed for 57 days after administration
  To evaluate the exploratory PD profile following single administration of YH35324
Change in serum soluble FcƐRI concentration | Change in serum soluble FcƐRI concentration will be observed for 57 days after administration
  To evaluate the exploratory PD profile following single administration of YH35324
Change in serum Mas-related G protein-coupled receptor-X2 (MRGPRX2) concentration | Change in serum Mas-related G protein-coupled receptor-X2 (MRGPRX2) concentration will be observed for 57 days after administration
  To evaluate the exploratory PD profile following single administration of YH35324
[Parts 1 and 2 only] Change in Basophil Histamine Release Assay (BHRA) | Change in Basophil Histamine Release Assay (BHRA) will be observed for 57 days after administration
  To evaluate the exploratory PD profile following single administration of YH35324
Change in the Urticaria Control Test (UCT) score | Change in the Urticaria Control Test (UCT) score will be observed for 57 days after administration
  To explore the clinical efficacy following single administration of YH35324
  * Urticaria Control Test score
  * minimum value: 0 / maximum value: 16
  * Higher scores mean a better outcome
Rate of Use of rescue medications | Use of rescue medications will be observed for 57 days after administration
  To explore the clinical efficacy following single administration of YH35324 for using rescue medications diary
[Parts 1 and 2 only] Change in weekly Hive Severity Score 7 (HSS7) | Change in weekly Hive Severity Score 7 (HSS7) will be observed for 57 days after administration
  To explore the clinical efficacy following single administration of YH35324
  * Hive Severity Score 7
  * minimum value: 0 / maximum value: 21
  * Higher scores mean a worse outcome
[Parts 1 and 2 only] Change in weekly Itch Severity Score 7 (ISS7) | Change in weekly Itch Severity Score 7 (ISS7) will be observed for 57 days after administration
  To explore the clinical efficacy following single administration of YH35324
  * Itch Severity Score 7
  * minimum value: 0 / maximum value: 21
  * Higher scores mean a worse outcome
[Parts 1 and 2 only] Change in weekly Urticaria Activity Score 7 (UAS7) | Change in weekly Urticaria Activity Score 7 (UAS7) will be observed for 57 days after administration
  To explore the clinical efficacy following single administration of YH35324
  * Urticaria Activity Score 7
  * minimum value: 0 / maximum value: 42
  * Higher scores mean a worse outcome
[Part 3 only] Change in Critical Temperature Thresholds (CTT) in response to the challenge test (TempTest® 4) | Change in Critical Temperature Thresholds (CTT) in response to the challenge test (TempTest® 4) will be observed for 57 days after administration
  To explore the clinical efficacy following single administration of YH35324
[Part 3 only] Change in the Peak Pruritus Numerical Rating Scale (PP-NRS) score after the challenge test (TempTest® 4) | Change in the Peak Pruritus Numerical Rating Scale (PP-NRS) score after the challenge test (TempTest® 4) will be observed for 57 days after administration
  To explore the clinical efficacy following single administration of YH35324
  * Peak Pruritus Numerical Rating Scale
  * minimum value: 0 / maximum value: 10
  * Higher scores mean a worse outcome
Incidence of serum anti-YH35324 antibodies | Incidence of serum anti-YH35324 antibodies will be observed for 57 days after administration
  To explore the immunogenicity following single administration of YH35324

CONTACTS AND LOCATIONS:
Overall Officials: Hae-Sim Park, Study Chair — Ajou University School of Medicine
Locations (9):
- South Korea (9):
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si, Gyeonggi-do
  - CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Dong-a University hospital, Busan
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including data dictionaries) that underline the results reported in study-related publications will be made available during the period beginning 1 year and ending 5 years after all trial primary and secondary endpoints were assessed. Only requests from researchers who provide a methodologically sound proposal will be reviewed and approved by the sponsor. The analysis type should be in accordance with aims in the proposal approved by the sponsor. Proposals should be directed to yjshim@yuhan.co.kr
  A summary of the study results will be posted in the publicly accessible database (i.e. clinicaltrials.gov) no later than 1 year after the study's primary completion date.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 1 year and ending 5 years after all trial endpoints were assessed
Access Criteria: Only requests from researchers who provide a methodologically sound proposal will be reviewed and approved by the sponsor. The analysis type should be in accordance with aims in the proposal approved by the sponsor. Proposals should be directed to yjshim@yuhan.co.kr